CLINICAL TRIAL: NCT01873417
Title: A Multicenter, Open-Label, Single-Arm Study of Gastrointestinal Tolerability in Patients With Relapsing Forms of Multiple Sclerosis Receiving Tecfidera™ (Dimethyl Fumarate) Delayed-release Capsules
Brief Title: Phase 4 Gastrointestinal Tolerability Study of Dimethyl Fumarate in Patients With Relapsing Forms of Multiple Sclerosis in the United States
Acronym: MANAGE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109MS403
Record Dates: First submitted 2013-05-09; First posted 2013-06-10 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Relapsing Forms of Multiple Sclerosis
MeSH Terms: interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dimethyl Fumarate (Experimental): 120 mg DMF twice daily (BID) for the first 7 days and 240 mg DMF BID thereafter for 12 weeks of treatment. Participants will be instructed to take the DMF dose with food (with a meal or within 1 hour after a meal).
  Interventions: Drug: BG00012 (DMF)

INTERVENTIONS:
Drug: BG00012 (DMF)
  Other Names: Tecfidera; DMF; dimethyl fumarate

SUMMARY:
The primary objective of this study is to evaluate the effect of symptomatic therapies on gastrointestinal (GI)-related events reported by participants with relapsing forms of multiple sclerosis (MS) initiating therapy with dimethyl fumarate (DMF) in the clinical practice setting.

The secondary objectives of this study are as follows:

* To evaluate GI-related events requiring symptomatic therapy and the role of those therapies over time in participants with relapsing forms of MS initiating therapy with DMF in the clinical practice setting.
* To evaluate GI-related events that lead to DMF discontinuation after the use of symptomatic therapy in participants with relapsing forms of MS initiating therapy with DMF in the clinical practice setting.

ELIGIBILITY:
Key Inclusion Criteria:

* Decision to treat with DMF must precede enrollment.
* Naïve to DMF or fumaric acid esters.
* Resides in the US and has a confirmed diagnosis of a relapsing form of MS.
* Satisfies the approved therapeutic indication(s) for DMF.

Key Exclusion Criteria:

* Inability to comply with study requirements or, at the discretion of the Investigator, is deemed unsuitable for study participation.
* History of significant GI disease, chronic use of GI symptomatic therapy, active malignancies.
* Is participating in any other interventional clinical trial.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (36):
- United States (36):
  - Research Site, Cullman, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Fullerton, California
  - Research Site, Newport Beach, California
  - Research Site, Pasadena, California
  - Research Site, Englewood, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Maitland, Florida
  - Research Site, Naples, Florida
  - Research Site, North Palm Beach, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Milford, Massachusetts
  - Research Site, Golden Valley, Minnesota
  - Research Site, Patchogue, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Portland, Oregon
  - Research Site, Monroeville, Pennsylvania
  - Research Site, Cordova, Tennessee
  - Research Site, Franklin, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Round Rock, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin

REFERENCES:
- [Background] Fox EJ, Vasquez A, Grainger W, Ma TS, von Hehn C, Walsh J, Li J, Zambrano J. Gastrointestinal Tolerability of Delayed-Release Dimethyl Fumarate in a Multicenter, Open-Label Study of Patients with Relapsing Forms of Multiple Sclerosis (MANAGE). Int J MS Care. 2016 Jan-Feb;18(1):9-18. doi: 10.7224/1537-2073.2014-101. PMID 26917993

RESULTS

PARTICIPANT FLOW:
Groups:
- Dimethyl Fumarate: 120 mg dimethyl fumarate (DMF) twice daily (BID) for the first 7 days and 240 mg DMF BID thereafter for 12 weeks of treatment. Participants were instructed to take the DMF dose with food (with a meal or within 1 hour after a meal).
Period: Overall Study
Arm/Group | Dimethyl Fumarate
Started | 237
Safety Population | 233 (Participants who received at least 1 dose of dimethyl fumarate (DMF), recorded in diary data.)
Completed | 202
Not Completed | 35
Not completed — Did Not Receive Any Study Drug | 4
Not completed — Adverse Event | 24
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: Safety Population (participants who received at least 1 dose of DMF, recorded in diary data)
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: Worst Severity Score of Overall Gastrointestinal (GI) Events, Modified Overall GI Symptom Scale (MOGISS)
Description: Severity of GI-related events in DMF-treated participants using the MOGISS to measure GI symptoms, based on a 0- to 10-point scale, with 0 representing absence of symptoms and 10 representing the most severe symptoms.
Time Frame: 12 Weeks
Population: Evaluable participants (treated participants who utilized symptomatic therapy during the overall treatment period [12 weeks]).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 128
units on a scale | 4.8 (2.34)

2. Primary Outcome: Worst Severity Score of Overall GI Events, Modified Acute Gl Symptom Scale
Description: Severity of GI-related events in DMF-treated participants using the MAGISS to measure GI symptoms, based on a 0- to 10-point scale, with 0 representing absence of symptoms and 10 representing the most severe symptoms.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 128
units on a scale | 4.7 (2.13)

3. Primary Outcome: Percentage of DMF-treated Participants Who Reported GI-related Symptoms and Who Utilized Symptomatic Therapy
Description: Percentage of participants reporting GI symptoms on the MOGISS, by those who utilized symptomatic therapy.
Time Frame: 12 Weeks
Population: Safety Population (participants who received at least 1 dose of DMF, recorded in diary data)
Measure: Number; unit: percentage of participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 233
percentage of participants | 54.1

4. Primary Outcome: Duration of GI-related Episodes in DMF-treated Participants
Description: In participants who took symptomatic therapy, the median duration of acute GI episodes (in hours) was summarized for the overall treatment period, by symptom (nausea, diarrhea, lower abdominal pain, upper abdominal pain, vomiting, indigestion, constipation, bloating, and flatulence). Table only includes the symptom duration for those symptoms with start and stop times entered in the eDiary (evaluable GI episodes), based on the MAGISS.
Time Frame: 12 Weeks
Population: Evaluable participants (treated participants who utilized symptomatic therapy during the overall treatment period [12 weeks]); n=number of participants with evaluable GI symptom specified.
Measure: Median (Full Range); unit: hours
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 128
hours
  Nausea; n=88 | 2.0 (1.81) [0.0 to 8.8]
  Diarrhea; n=78 | 1.6 [0.0 to 11.0]
  Lower Abdominal Pain; n=67 | 2.0 [0.0 to 8.0]
  Upper Abdominal Pain; n=66 | 1.8 [0.1 to 9.5]
  Vomiting; n=27 | 0.4 [0.0 to 8.0]
  Indigestion; n=52 | 1.9 [0.0 to 11.0]
  Constipation; n=7 | 6.0 [0.0 to 23.0]
  Bloating; n=41 | 3.0 [0.0 to 12.7]
  Flatulence; n=68 | 2.1 [0.2 to 12.7]

5. Secondary Outcome: Percentage of DMF-treated Participants Who Required GI Symptomatic Therapy
Description: Percentage of participants reporting that they required GI symptomatic therapy, based on the MOGISS.
Time Frame: 12 Weeks
Population: Safety Population (participants who received at least 1 dose of DMF, recorded in diary data)
Measure: Number; unit: percentage of participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 233
percentage of participants | 54.1

6. Secondary Outcome: Participants' Use of Symptomatic Therapy, by Type and Category
Description: The symptomatic therapies used by DMF-treated participants were self-reported by type and category. Each participant may have taken more than one symptomatic therapy type but was counted only once within each therapy category. Acetylsalicylic acid (ASA) is abbreviated in the table.
Time Frame: 12 Weeks
Population: Safety Population (participants who received at least 1 dose of DMF, recorded in diary data)
Measure: Number; unit: participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 233
participants
  Category: Antacid | 57
  Therapy: Calcium carbonate | 50
  Therapy: Magnesium (Mg) hydroxide | 4
  Therapy: Aluminum (Al) hydroxide | 1
  Therapy: Al hydroxide, Mg hydroxide, simethicone | 3
  Therapy: ASA, citric acid, sodium bicarbonate | 2
  Therapy: Generic anatacid | 1
  Therapy: Nauzene | 1
  Therapy: Sucralfate | 1
  Category: Antisecretory/antimicrobial | 49
  Therapy: Bismuth subsalicylate | 49
  Category: Anti-acid production | 43
  Therapy: Omeprazole | 18
  Therapy: Ranitidine | 15
  Therapy: Famotidine | 14
  Therapy: Lansoprazole | 10
  Therapy: Pantoprazole | 3
  Therapy: Cimetidine | 1
  Category: Anti-bloating/anti-constipation agent | 33
  Therapy: Simethicone | 29
  Therapy: Docusate | 5
  Therapy: Alpha-galactosidase | 1
  Therapy: Enema | 1
  Category: Antidiarrheal (anti-peristaltic) | 32
  Therapy: Loperamide | 29
  Therapy: Diphenoxylate | 3
  Therapy: Dicyclomine | 2
  Category: Anti-emetic (central) | 18
  Therapy: Ondansetron | 8
  Therapy: Promethazine | 7
  Therapy: Dimenhydrinate | 3
  Therapy: Tetrahydrocannabinol | 1
  Category: Laxative, fiber/probiotic | 10
  Therapy: Generic laxative | 5
  Therapy: Psyllium fiber | 3
  Therapy: Culturelle | 2
  Category: Laxative, hygroscopic/osmotic | 10
  Therapy: Polyethylene glycol | 4
  Therapy: Phosphorated carbohydrate solution | 3
  Therapy: Sennosides | 2
  Therapy: Osmotic | 1
  Category: Laxative, prokinetic | 7
  Therapy: Bisacodyl | 7
  Category:Analgesic (nonsteroidal antiinflammatory) | 5
  Therapy: Ibuprofen | 3
  Therapy: Naproxen | 2
  Therapy: ASA | 1
  Category: Anti-allergic | 3
  Therapy: Montelukast | 2
  Therapy: Diphenhydramine | 1
  Category: Anti-emetic (pro-kinetic) | 3
  Therapy: Metoclopramide | 3
  Category: Analgesic | 2
  Therapy: Acetaminophen | 2
  Category: No treatment type recorded | 1
  Therapy: Not available | 1

7. Secondary Outcome: Summary of Use and Days on Symptomatic Therapy, by Category
Description: The total duration (in days) of use of each symptomatic therapy by participants as a result of GI symptoms experienced by DMF-treated participants is presented. If a participant had multiple different therapies on the same day, the days on symptomatic therapy was calculated as 1 day in the 'All Therapies' category.
Time Frame: 12 Weeks
Population: Evaluable participants (treated participants who utilized symptomatic therapy during the overall treatment period [12 weeks]). n= number of participants using the therapy specified.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 128
days
  All therapies; n=128 | 10.4 (13.46)
  Antacid; n=57 | 5.9 (10.77)
  Antisecretory/antimicrobial; n=49 | 6.3 (12.34)
  Anti-acid production; n=43 | 9.0 (11.16)
  Anti-bloating/anti-constipation agent; n=33 | 5.9 (10.86)
  Anti-diarrheal (anti-peristaltic); n=32 | 3.9 (3.88)
  Anti-emetic (central); n=18 | 2.9 (2.00)
  Laxative, fiber/probiotic; n=10 | 5.0 (5.64)
  Laxative, hygroscopic/osmotic; n=10 | 3.7 (3.06)
  Laxative, prokinetic; n=7 | 1.6 (0.79)
  Analgesic (nonsteroidal antiinflammatory); n=5 | 4.6 (7.50)
  Anti-allergic; n=3 | 12.0 (9.85)
  Anti-emetic; n=3 | 9.7 (12.42)
  Analgesic; n=2 | 4.5 (4.95)
  No treatment type recorded; n=1 | 1.0 (NA) — only 1 participant analyzed

8. Secondary Outcome: Number of DMF-treated Participants Who Discontinued DMF Due to GI-related Events Requiring Symptomatic Therapy
Description: The last symptomatic therapy prior to last dose of study medication was used to summarize the number of participants who discontinued DMF due to GI-related events. Participants may have taken more than one symptomatic therapy but are counted only once in the 'All Therapies' category.
Time Frame: 12 Weeks
Population: Safety Population (participants who received at least 1 dose of DMF, recorded in diary data)
Measure: Number; unit: participants
Arm/Group | Dimethyl Fumarate
Number analyzed (Participants) | 233
participants
  All therapies | 13
  Anti-acid production | 10
  Antacid | 6
  Antisecretory/antimicrobial | 6
  Anti-diarrheal (anti-peristaltic) | 5
  Anti-emetic (central) | 5
  Anti-emetic (prokinetic) | 2
  Laxative, fiber/probiotic | 1
  Laxative, prokinetic | 1

ADVERSE EVENTS:
Time Frame: All serious adverse events (SAEs) from time of signed/dated informed consent through 12 weeks of treatment plus 4 weeks (± 5 days) post last dose.
Description: Non-serious adverse events (other than GI-related events and events resulting in discontinuation of the study drug or withdrawal from the study) were not collected in this study, per protocol.
Arm/Group | Dimethyl Fumarate
Serious Adverse Events (participants affected / at risk) | 7/233
Other Adverse Events (participants affected / at risk) | 0/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dimethyl Fumarate (N=233)
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Salivary Gland Calculus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Sudden Cardiac Death (General disorders) | 1
Troponin Increased (Investigations) | 1
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1
Confusional State (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.